CLINICAL TRIAL: NCT01436955
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Multiple Dose Study to Investigate Safety and Tolerability of RG1662 in Individuals With Down Syndrome
Brief Title: A Study of RG1662 in Individuals With Down Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP25543
Record Dates: First submitted 2011-08-18; First posted 2011-09-20 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: RG1662
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — multiple oral doses
  Arms: B
Drug: RG1662 — Cohorts receiving multiple oral doses
  Arms: A

SUMMARY:
This multi-center, randomized double-blind, placebo-controlled study will assess the safety and tolerability of RG1662 in individuals with Down Syndrome. Eligible subjects will be randomized in cohorts to receive either multiple oral doses of RG1662 or placebo. Anticipated time on study treatment is 38 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals, 18 to 30 years of age, with diagnosis of Down Syndrome (confirmed by karyotype)
* Males and non-pregnant non-lactating females
* Parent or legal guardian/representative and caregiver willing to give written informed consent
* Subject willing and assenting or consenting to participate

Exclusion Criteria:

* Major depressive disorder not adequately controlled by a selective serotonin reuptake inhibitor or a serotonin norepinephrine reuptake inhibitor
* Subjects meeting clinical diagnostic criteria for autistic spectrum disorder, attention deficit or hyperactivity disorder unlikely to cooperate and take part successfully in the study assessments
* Subjects with other primary psychiatric diagnosis
* Subjects with evidence or meeting clinical diagnosis of dementia
* Subjects with personal history of cardiac abnormalities; patients that have previously undergone congenital heart surgery can be enrolled provided they have no residual complication requiring intervention (e.g. pace maker)
* Subjects with clinically significant obstructive pulmonary disease or asthma that is not adequately treated (oral steroids are not allowed)
* Subjects with thyroid dysfunction that is not adequately controlled and stabilized on treatment for at least 8 weeks
* Subjects with sustained elevated supine blood pressure (SBP/DBP) at rest exceeding 140/90 mmHg or notable resting tachycardia (mean HR > 60 bpm) or blood pressure below 90/40 mmHg
* Subjects who have taken any other investigational medications within 3 months
* Body mass index (BMI) > 40 kg/m2

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 16 weeks

SECONDARY OUTCOMES:
Neurocognitive assessment: CANTAB (Computerized battery for assessing motor practice, reaction time and memory)/standard cognitive tests | 5-6 weeks
Pharmacokinetics: Serum concentration/area under the concentration-time curve (AUC) | 5-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- United States (8):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - La Jolla, California
  - Aurora, Colorado
  - Decatur, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Durham, North Carolina
- London, United Kingdom